CLINICAL TRIAL: NCT06452238
Title: External Oblique Intercostal Plane Block Versus Ultrasound Guided Transversus Abdominis Plane Block for Postoperative Analgesia in Adult Patients Undergoing Open Nephrectomy
Brief Title: External Oblique Intercostal Plane Block Versus Transversus Abdominis Plane Block for Postoperative Analgesia in Adult Patients Undergoing Open Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR639/4/24
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: External Oblique Intercostal Plane Block; Transversus Abdominis Plane Block; Postoperative Analgesia; Nephrectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Oblique Intercostal Plane Block (Experimental): Patients will receive external oblique intercostal plane block .
  Interventions: Other: External Oblique Intercostal Plane Block
- Transversus Abdominis Plane Block (Experimental): Patients will receive ultrasound guided transversus abdominis plane block.
  Interventions: Other: Transversus Abdominis Plane Block

INTERVENTIONS:
Other: External Oblique Intercostal Plane Block — Patients will receive external oblique intercostal plane block .
  Arms: External Oblique Intercostal Plane Block
Other: Transversus Abdominis Plane Block — Patients will receive ultrasound-guided transversus abdominis plane block.
  Arms: Transversus Abdominis Plane Block

SUMMARY:
The aim of this study is to compare external oblique intercostal plane (EOIP) block and ultrasound guided transversus abdominis plane (TAP) Block for postoperative analgesia in adult patients undergoing open nephrectomy.

DETAILED DESCRIPTION:
Patients undergoing nephrectomy have a high incidence of postoperative pain despite the use of modern laparoscopic surgical techniques. In the postoperative period, these patients are often treated with patient-controlled opioids, epidural analgesia, or both.

Ultrasound-guided transversus abdominis plane (TAP) block is a relatively new technique to infiltrate regional anesthesia in which local routine anesthetics are injected between the internal oblique and transverse abdominal muscles. Studies have confirmed that ultrasound-guided (USG) transversus abdominis plane (TAP) block is an effective method of analgesia for upper abdominal surgeries, lower abdominal surgeries, and kidney transplantation, with minimal side effects.

External oblique intercostal plane block (EOIPB) has been reported by Elsharkawy et al. in 2021 as a significant modification of fascial plane blocks in that it may engage the upper lateral abdominal walls consistently. In comparison to quadratus lumborum block (QLB) and erector spinae plane block (ESPB) , The advantage of EOIPB is that it may be performed with the patient supine. Furthermore, in comparison to serratus intercostal plane block (SIPB), it generates more extensive analgesic effects throughout the whole midline of the abdomen .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for open nephrectomy.

Exclusion Criteria:

* Bleeding disorders.
* Skin lesions or infection at the site of proposed needle insertion.
* Allergy to local anesthetics.
* Neurological disorders.
* Drug abuse.
* BMI > 30 kg/m2.
* Pregnancy.
* Diabetic neuropathy.
* Severe cardiovascular problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Total pethidine consumption in the 1st 24hr | 24 hours postoperatively
  A standardized analgesic regimen will be prescribed in the postoperative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia. Rescue analgesia of pethidine will be given as 2 mg bolus if the Numerical Rating Scale (NRS) > 3 to be repeated after 30 min if pain persists until the Numerical Rating Scale (NRS) < 4. NRS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Time to the 1st rescue analgesia. | 24 hours postoperatively
  A standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia. Rescue analgesia of pethidine will be given as 2 mg bolus if the Numerical Rating Scale (NRS) > 3 to be repeated after 30 min if pain persists until the Numerical Rating Scale (NRS) < 4. NRS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.
  It will be measured from the end of surgery to first dose of pethidine administrated.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.
Mean arterial pressure | Every 15 minutes till the end of surgery
  It will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Heart rate | Every 15 minutes till the end of surgery
  It will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author